CLINICAL TRIAL: NCT00470067
Title: A Multi-center Phase II Study of Doxil®/Carboplatin in Patients With Advanced or Recurrent Endometrial Carcinoma
Brief Title: Doxorubicin Hydrochloride Liposome and Carboplatin in Treating Patients With Recurrent, Stage III, or Stage IV Primary Endometrial Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to low accrual
Sponsor: Roswell Park Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000543389; RPCI-I-68005
Record Dates: First submitted 2007-05-03; First posted 2007-05-07 (Estimated); Results first posted 2014-08-22 (Estimated); Last update posted 2014-08-22 (Estimated); Status verified 2014-08

CONDITIONS: Endometrial Cancer
Keywords: recurrent endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Doxorubicin and carboplatin (Experimental): Patients receive doxorubicin hydrochloride liposome IV over 1 hour on day 1 and carboplatin IV over 30 minutes on day 1
  Interventions: Drug: carboplatin; Drug: pegylated liposomal doxorubicin hydrochloride

INTERVENTIONS:
Drug: carboplatin — IV
Drug: pegylated liposomal doxorubicin hydrochloride — IV

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as doxorubicin hydrochloride liposome and carboplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving doxorubicin hydrochloride liposome together with carboplatin works in treating patients with recurrent, stage III, or stage IV primary endometrial cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Estimate the response rate in patients with recurrent or stage III or IV primary endometrial carcinoma treated with doxorubicin hydrochloride liposome and carboplatin.

Secondary

* Determine progression-free survival of patients treated with this regimen.
* Determine overall survival of patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive doxorubicin hydrochloride liposome IV over 1 hour on day 1 and carboplatin IV over 30 minutes on day 1. Treatment repeats every 28 days for up to 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed at 6 months and then every 3 months thereafter.

PROJECTED ACCRUAL: A total of 37 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed primary endometrial carcinoma meeting 1 of the following criteria:

  * Stage III or IV disease according to FIGO staging criteria
  * Recurrent disease that is considered incurable
* Measurable disease

  * A lesion within a previously irradiated field is acceptable as measurable disease only if there has been clear progression since completion of radiotherapy

PATIENT CHARACTERISTICS:

* GOG performance status 0-2
* Absolute neutrophil count ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* Creatinine < 2.5 mg/dL OR creatinine clearance ≥ 60 mL/min
* ALT and AST ≤ 1.5 times upper limit of normal (ULN) (3 times ULN in the presence of liver metastases)
* Alkaline phosphatase ≤ 1.5 times ULN (3 times ULN in the presence of liver metastases)
* Total bilirubin ≤ 1.5 times ULN (3 times ULN in the presence of liver metastases)
* Not pregnant or nursing
* Left ventricular ejection fraction (LVEF) ≥ 50% by MUGA scan or ECHO
* No history of severe hypersensitivity reaction to doxorubicin hydrochloride liposome
* No other invasive malignancy (i.e., breast cancer) within the past 5 years except nonmelanoma skin cancer
* No cardiac disease, including any of the following:

  * Myocardial infarction within the past 6 months
  * NYHA class II-IV heart failure
  * Uncontrolled angina
  * Severe uncontrolled ventricular arrhythmias
  * Clinically significant pericardial disease
  * Acute ischemic or active conduction system abnormalities by ECHO

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy
* No prior cancer therapy that would contraindicate study treatment
* No concurrent investigational agents

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2007-02; Primary Completion 2008-05 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shashikant B. Lele, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (1):
- Roswell Park Cancer Institute, Buffalo, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doxorubicin and Carboplatin
Started | 9
Completed | 2
Not Completed | 7
Not completed — Death | 1
Not completed — Disease Progression | 6

BASELINE CHARACTERISTICS:
Population: All treated and eligible patients
Arm/Group | Doxorubicin and Carboplatin
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.9 (8.04)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Response (Complete and Partial)
Description: Response Rate
Time Frame: Every 28 days
Population: Due to the study's early termination and inadequate number of patients, no patients were analyzed.
Arm/Group | Doxorubicin and Carboplatin
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Doxorubicin and Carboplatin
Serious Adverse Events (participants affected / at risk) | 2/9
Other Adverse Events (participants affected / at risk) | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin and Carboplatin (N=9)
Neutropenia (Blood and lymphatic system disorders) | 1 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (2)
Death (General disorders) | 1 (2)
Infection (Infections and infestations) | 1 (2)
Septic shock (Infections and infestations) | 1 (2)
Blood creatinine increased (Investigations) | 1 (2)
White blood cell count decreased (Investigations) | 1 (2)
Syncope (Nervous system disorders) | 1 (2)
Renal failure (Renal and urinary disorders) | 2 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Doxorubicin and Carboplatin (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 (4)
Ear pain (Ear and labyrinth disorders) | 1 (2)
Tinnitus (Ear and labyrinth disorders) | 1 (2)
Abdominal pain (Gastrointestinal disorders) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (4)
Diarrhoea (Gastrointestinal disorders) | 2 (4)
Nausea (Gastrointestinal disorders) | 1 (2)
Asthenia (General disorders) | 2 (4)
Fatigue (General disorders) | 5 (10)
Oedema peripheral (General disorders) | 3 (6)
Pyrexia (General disorders) | 2 (6)
Herpes simplex (Infections and infestations) | 1 (2)
Wound infection (Infections and infestations) | 1 (2)
Blood alkaline phosphatase (Investigations) | 1 (2)
Blood creatine increased (Investigations) | 1 (2)
Blood creatinine increased (Investigations) | 1 (4)
Blood urea increased (Investigations) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 2 (4)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Hypercalcaemia (Metabolism and nutrition disorders) | 2 (4)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 (2)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (8)
Hyperkalaemia (Metabolism and nutrition disorders) | 2 (4)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2)
Neuropathy peripheral (Nervous system disorders) | 1 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (2)
Anxiety (Psychiatric disorders) | 1 (2)
Vaginal burning sensation (Reproductive system and breast disorders) | 1 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Dermatitis (Skin and subcutaneous tissue disorders) | 1 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (2)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (2)
Stent placement (Surgical and medical procedures) | 1 (2)
Deep vein thrombosis (Vascular disorders) | 1 (2)
Hypertension (Vascular disorders) | 1 (2)

LIMITATIONS AND CAVEATS:
Due to the study's early termination and inadequate number of patients, no patients were analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes